CLINICAL TRIAL: NCT04510285
Title: A Single-Arm Pilot Study of Adjuvant Pembrolizumab Plus Trastuzumab in HER2+ Esophagogastric Tumors With Persistent Circulating Tumor DNA Following Curative Resection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-158
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Esophagogastric Tumors; Gastric Cancer; Gastric Tumor; Esophageal Cancer; Esophageal Neoplasms; Esophageal Tumor; GastroEsophageal Cancer; Gastroesophageal Junction Adenocarcinoma; Gastroesophageal Junction Tumor; Gastroesophageal Junction Cancer
Keywords: Esophagogastric Tumors; Esophagogastric Cancers; Gastric Cancer; Esophageal Cancer; Gastroesophageal Junction Cancer; GEJ Tumor; Pembrolizumab; Trastuzumab; 20-158; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Trastuzumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a single arm pilot study of adjuvant pembrolizumab + trastuzumab.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trastuzumab and Pembrolizumab (Experimental): Trastuzumab will be administered on an every 3 week dosing schedule, with initial loading dose of 8 mg/kg as a 90 minute infusion, followed by trastuzumab 6 mg/kg every 3 weeks.
  The planned dose of pembrolizumab for this study is 200 mg every 3 weeks.
  Interventions: Drug: Trastuzumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab (8mg/kg loading dose; 6mg/kg maintenance) will be administered on day 1 of each 3-week dosing cycle (21 days).
Drug: Pembrolizumab — Pembrolizumab 200 mg IV will be administered on day 1 of each 3-week dosing cycle (21 days).

SUMMARY:
The purpose of this study is to find out whether treatment with trastuzumab combined with pembrolizumab will improve the clearance of tumor DNA from participants' bodies after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* ECOG performance status 0-2.
* Sign informed consent within 8 months after curative surgery and completion of standard of care perioperative and/or adjuvant therapy.
* HER2+ esophageal, GEJ, or gastric adenocarcinoma biopsy or resection specimen as defined by local HER2 IHC3+ or IHC 2+/FISH>2.0 expression.
* Must have genetic testing of DNA from primary tumor for somatic genomic alterations across a minimum of 50 genes.
* Must have undergone a complete curative surgical resection (R0).
* Must have completed standard of care (SOC) surgery, neoadjuvant or adjuvant therapy
* CtDNA will be tested at a minimum of four weeks after completion of surgery and standard perioperative and/or adjuvant therapy. To be eligible for trastuzumab/pembrolizumab or trastuzumab therapy, the patients must have positive ctDNA (as defined in section 7.0) within 8 months after completion of appropriate standard of care therapy (surgery, chemotherapy, radiation as appropriate). For all patients, if the initial ctDNA has a negative result, ctDNA can be re-tested 4 weeks later, within 9 months of completion of standard therapy.
* Demonstrate adequate organ function as defined in Table 1.

Hematological Absolute neutrophil Count (ANC): ≥ 1,500 /mcL Platelets: ≥ 100,000 /mcL Hemoglobin: ≥ 9 g/dL

Renal Serum creatinine ≤ 1.5 X upper limit of normal (ULN)

Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN. Except patients with Gilbert's disease (≤ 3 x ULN) AST and ALT ≤ 2.5 X ULN Albumin ≥ 3 mg/dL

Exclusion Criteria:

* Patients who have not recovered from serious adverse events (as determined by treating MD) related to surgery.
* Presence of metastatic or recurrent disease.
* Had R1 (microscopic residual tumor) or R2 resection (macroscopic residual tumor at resection margin).
* Left ventricular ejection fraction <50% within 1 month of screening by MUGA or echocardiogram.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., dexamethasone containing antiemetic regimen or steroids as CT scan contrast premedication) may be enrolled.
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  ° Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-CTLA-4 agent.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

  ° Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Is unwilling to give written informed consent, unwilling to participate, or unable to comply with the protocol for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Y Janjigian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab and Pembrolizumab: Trastuzumab will be administered on an every 3 week dosing schedule, with initial loading dose of 8 mg/kg as a 90 minute infusion, followed by trastuzumab 6 mg/kg every 3 weeks.
  The planned dose of pembrolizumab for this study is 200 mg every 3 weeks.
  Trastuzumab: Trastuzumab (8mg/kg loading dose; 6mg/kg maintenance) will be administered on day 1 of each 3-week dosing cycle (21 days).
  Pembrolizumab: Pembrolizumab 200 mg IV will be administered on day 1 of each 3-week dosing cycle (21 days).
Period: Overall Study
Arm/Group | Trastuzumab and Pembrolizumab
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab and Pembrolizumab
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 86 [86 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of ctDNA Clearance at 6 Months
Description: The primary endpoint of the study is the proportion of patients with ctDNA clearance at 6 months with trastuzumab/pembrolizumab or trastuzumab/placebo in patients with HER2+ esophagogastric cancer with persistent ctDNA despite curative surgery and standard perioperative/adjuvant therapy.
  CtDNA clearance is the conversion of detectable to undetectable ctDNA
Time Frame: 6 months
Population: N/A - data were not collected because the one participant accrued to the study died prematurely due to a treatment unrelated infection
Arm/Group | Trastuzumab and Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Trastuzumab and Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Pembrolizumab (N=1)
Sepsis (Infections and infestations) | 1
Death NOS (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Pembrolizumab (N=1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT04510285/Prot_SAP_000.pdf